CLINICAL TRIAL: NCT03081052
Title: Inhaled Selective Pulmonary Vasodilators for Advanced Heart Failure Therapies and Lung Transplantation Outcomes
Acronym: INSPIRE-FLO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Pro00078035
Record Dates: First submitted 2017-03-08; First posted 2017-03-15 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Heart Transplant Surgery; Lung Transplant Surgery
Keywords: Heart and Lung transplantation surgery; Pulmonary vasodilation therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lung transplant with iNO (Active Comparator)
  Interventions: Drug: iNO
- Lung transplant with iEPO (Active Comparator)
  Interventions: Drug: iEPO
- Heart transplant & LVAD implantation with iNO (Active Comparator)
  Interventions: Drug: iNO
- Heart transplant & LVAD implantation with iEPO (Active Comparator)
  Interventions: Drug: iEPO

INTERVENTIONS:
Drug: iNO — Subject will receive inhaled Nitric Oxide in this intervention
  Other Names: Inhaled Nitric Oxide
  Arms: Heart transplant & LVAD implantation with iNO; Lung transplant with iNO
Drug: iEPO — Subject will receive inhaled Epoprostrenol in this intervention
  Other Names: Inhaled Epoprostrenol
  Arms: Heart transplant & LVAD implantation with iEPO; Lung transplant with iEPO

SUMMARY:
1. to conduct a clinical investigation to determine if inhaled epoprostenol (Veletri®, iEPO) and inhaled nitric oxide (iNO) will have similar impact on outcomes in adult patients undergoing durable LVAD placement, heart transplantation, or lung transplantation 2. to conduct a cost-capture analysis on the expense each drug incurs per patient.

DETAILED DESCRIPTION:
In adult cardiothoracic surgical patients, iNO is used to treat precapillary pulmonary hypertension (PH), right-sided heart failure (RHF), and ventilation-to-perfusion (V:Q) mismatch. Adult patients who undergo durable LVAD implantation (e.g. Heartware®, Heartmate 2®, or Heartmate 3®), cardiac transplantation for HFrEF, or those that have endured lung transplantation as a result of end-stage lung disease, compose the largest subpopulation which receives iPVD therapy at Duke University Hospital. iEPO may display an equivalent efficacy profile to iNO for pulmonary vasodilation and oxygenation and have a similar impact on clinical outcomes.

Subjects undergoing LVAD placement or heart transplantation (N=224) or lung transplantation (N=200) will be prospectively enrolled over a three-year period (one-year for follow-up). Patients will be randomly assigned 1:1 according to stratified randomization blocking either iNO or iEPO. Additional study procedures will involve data collection, blood, and tissue sampling.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplantation
* LVAD placement
* Lung Transplantation

Exclusion Criteria:

* Combined Organ Transplantation
* Age < 18 years old
* Pregnancy
* Known allergy to prostaglandin (rare)
* Refusal of blood products due to personal or religious preference
* Subject is enrolled in another study protocol, which does not allow randomization of PVD therapy
* Heart transplant or durable LVAD recipients with adult congenital heart disease (CHD)

  o Caveat: Does NOT meet exclusion criteria if the scheduled heart transplant or LVAD implantation is due to heart failure from a previous heart transplantation related to CHD, performed more than 90 days previous to the date of trial enrollment
* Heart transplant recipients diagnosed with Arrythmogenic Right Ventricular Cardiomyopathy
* Heart transplant recipients diagnosed with Acute Cardiac Allograft Rejection after a previous heart transplantation.
* Heart transplant or durable LVAD recipients with preoperative RVAD for right heart failure
* Patient is scheduled to undergo lung transplantation but has undergone heart transplantation in the previous 90 days
* Patient is scheduled to undergo durable LVAD implantation but has undergone heart transplantation in the previous 90 days
* Patient is scheduled to undergo heart transplantation but has undergone lung transplantation in the previous 90 days
* Patients with preoperative Venovenous ECMO as a bridge to lung transplantation
* Heart transplant or durable LVAD recipients with preoperative RVAD for right heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2017-05-04 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2021-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kamrouz Ghadimi, MD, Principal Investigator — Duke Health
Locations (1):
- Duke Health, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghadimi K, Cappiello JL, Wright MC, Levy JH, Bryner BS, DeVore AD, Schroder JN, Patel CB, Rajagopal S, Shah SH, Milano CA; INSPIRE-FLO Investigators. Inhaled Epoprostenol Compared With Nitric Oxide for Right Ventricular Support After Major Cardiac Surgery. Circulation. 2023 Oct 24;148(17):1316-1329. doi: 10.1161/CIRCULATIONAHA.122.062464. Epub 2023 Jul 4. PMID 37401479
- [Derived] Ghadimi K, Cappiello J, Cooter-Wright M, Haney JC, Reynolds JM, Bottiger BA, Klapper JA, Levy JH, Hartwig MG; INSPIRE-FLO Investigators. Inhaled Pulmonary Vasodilator Therapy in Adult Lung Transplant: A Randomized Clinical Trial. JAMA Surg. 2022 Jan 1;157(1):e215856. doi: 10.1001/jamasurg.2021.5856. Epub 2022 Jan 12. PMID 34787647

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 519 participants were randomized, but 87 of those were unable to undergo surgery on protocol. 432 participants started the study (i.e., underwent surgery on protocol).
Period: Overall Study
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Started (Since these agents are standard of care at our institution for these operations, and either agent could be used outside of the study, participants were included in the analysis if they: 1. Did not die while awaiting surgery 2. Did not develop changes to enrollment criteria in the duration between consent and operation. 3. Was not withdrawn from study by physician before surgery) | 98 | 103 | 111 | 120
Completed (The number of patients who completed primary outcome follow-up) | 98 | 103 | 111 | 120
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients who were consented and randomized, but excluded or withdrawn prior to surgery and treatment are not included in this cohort description. No participant data was retained after patient exclusion or withdrawal prior to surgery and treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO | Total
Number analyzed (Participants) | 98 | 103 | 111 | 120 | 432
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [54 to 68] | 64 [51 to 69] | 59 [50 to 65] | 58 [48 to 65] | 60 [50 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 33 | 25 | 35 | 132
  Male | 59 | 70 | 86 | 85 | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 1 | 9
  Not Hispanic or Latino | 92 | 96 | 107 | 116 | 411
  Unknown or Not Reported | 4 | 4 | 1 | 3 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 9 | 44 | 47 | 112
  White | 83 | 91 | 66 | 72 | 312
  More than one race | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 Primary Graft Dysfunction (PGD) for Lung Transplant Subjects
Description: This is defined by the International Society of Heart and Lung Transplantation (ISHLT) as severe hypoxemia with a PaO2-to-FiO2 ratio < 200 or the presence of venovenous extracorporeal membrane oxygenation (VV ECMO) at a time-point within the first 72 hours after lung transplantation.
Time Frame: Up to 72 hours
Population: Only applicable to lung transplant patients on protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO
Number analyzed (Participants) | 98 | 103
Participants | 39 | 46
Statistical Analysis 1: Comparison: Lung Transplant With iNO vs Lung Transplant With iEPO; Test type: Equivalence — We estimated sample size based on equivalence test of the incidence rates of a binary outcome (e.g. PGD grade 3 (PGD-3)) of two treatment groups as an illustration. Assuming the incidence rate of PGD-3 under iEPO treatment is 0.30 and acceptable margin of the equivalence is ± 0.19, we will need 200 lung transplant patients to have 80% power to detect an actual difference at α=0.05 between two treatment group under this margin; p = 0.019, two one sided test p-value; Risk Difference (RD) = 0.049, 90% CI 2-sided [-0.064 to 0.162]

2. Primary Outcome: Number of Participants With Moderate or Severe RV Failure for the LVAD Implantation Subjects and Severe RV Failure for Heart Transplantation Subjects
Description: This is defined by the Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) score of moderate or severe right-heart failure for LVADS, and by the incidence of an RVAD placement or ECMO for RHF for heart transplants.
Time Frame: up to approximately 21 days after LVAD placement, up to approximately 30 days after heart transplantation
Population: Only applicable to heart transplant and LVAD implantation cohort that were treated on protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 111 | 120
Participants | 25 | 30
Statistical Analysis 1: Comparison: Heart Transplant & LVAD Implantation With iNO vs Heart Transplant & LVAD Implantation With iEPO; Test type: Non-Inferiority — We estimated sample size based on equivalence test of the incidence rates of a binary outcome of two treatment groups as an illustration. Assuming the incidence rate of moderate or severe RV failure under iEPO treatment is 0.113 and acceptable margin of the equivalence is ± 0.15, we will need 224 heart failure patients to have 80% power to detect an actual difference at α=0.05 between two treatment group under this margin; p = 0.012, two one-sided test p-value; Risk Difference (RD) = 0.025, 90% CI 2-sided [-0.066 to 0.116]

3. Secondary Outcome: Duration of Postoperative Mechanical Ventilation
Description: Length of time from intubation until patient is extubated
Time Frame: up to approximately 90 days after index surgery
Population: Among patients extubated, if patients transitioned directly from intubation to tracheostomy the duration of mechanical ventilation was censored at the time of tracheostomy placement
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Heart Transplant & LVAD Implantation With iNO: iNO: Subjects will receive inhaled Nitric Oxide in this intervention
- Heart Transplant & LVAD Implantation With iEPO: iEPO: Subjects will receive inhaled Epoprostrenol in this intervention
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 97 | 100 | 111 | 119
hours | 17 [12 to 47] | 18 [13 to 44] | 26 [12 to 48] | 24 [11 to 53]
Statistical Analysis 1: Comparison: Lung Transplant With iNO vs Lung Transplant With iEPO; Test type: Other; p = 0.747, Log Rank; Hodges-Lehmann Location Shift = 0, 95% CI 2-sided [-3 to 3]
Statistical Analysis 2: Comparison: Heart Transplant & LVAD Implantation With iNO vs Heart Transplant & LVAD Implantation With iEPO; Test type: Other; p = 0.638, Log Rank; Hodges-Lehmann Location Shift = 0, 95% CI 2-sided [-1 to 1]

4. Secondary Outcome: Per Patient Inhaled Pulmonary Vasodilator (iPVD) Cost
Description: Data reflects a per patient cost in dollars that has been scaled to a unit of measure relative to the cost per hour of drug and multiplied by the duration of iPVD administration. In our study, iNO cost 7 times that of iEPO per hour, hence for each patient this outcome value is the duration of iPVD administration multiplied by 7 if a patient is randomized to iNO or multiplied by 1 if randomized to iEPO.
Time Frame: up to approximately 30 days after index surgery
Measure: Mean (Standard Deviation); unit: relative cost units
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 98 | 103 | 111 | 120
relative cost units | 544 (513) | 70 (70) | 772 (554) | 114 (121)

5. Secondary Outcome: Length of ICU Stay
Description: Length of time from ICU admission from surgery until ICU discharge
Time Frame: up to approximately 90 days after index surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 98 | 103 | 111 | 120
days | 4 [2 to 10] | 4 [2 to 10] | 6 [4 to 11] | 6 [4 to 11]
Statistical Analysis 1: Comparison: Lung Transplant With iNO vs Lung Transplant With iEPO; Test type: Other; p = 0.453, log-linear regression; mean ratio = 1.19, 95% CI 2-sided [0.76 to 1.87]
Statistical Analysis 2: Comparison: Heart Transplant & LVAD Implantation With iNO vs Heart Transplant & LVAD Implantation With iEPO; Test type: Other; p = 0.816, log-linear regression; mean ratio = 0.94, 95% CI 2-sided [0.57 to 1.56]

6. Secondary Outcome: Length of Hospital Stay
Description: Length of time from surgery to hospital discharge
Time Frame: up to approximately 1 year after index surgery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 98 | 103 | 111 | 120
days | 23 [16 to 38] | 23 [15 to 38] | 16 [12 to 30] | 17 [11 to 28]
Statistical Analysis 1: Comparison: Lung Transplant With iNO vs Lung Transplant With iEPO; Test type: Other; p = 0.864, log-linear regression; mean ratio = 1.03, 95% CI 2-sided [0.75 to 1.41]
Statistical Analysis 2: Comparison: Heart Transplant & LVAD Implantation With iNO vs Heart Transplant & LVAD Implantation With iEPO; Test type: Other; p = 0.825, log-linear regression; mean ratio = 0.97, 95% CI 2-sided [0.73 to 1.28]

7. Secondary Outcome: Number of Participants With Acute Kidney Injury
Description: defined by Modified KDIGO-AKI definition:
  * Increase in Serum Creatinine (Cr) by ≥0.3mg/dL within 48 hours; or
  * Increase in Cr to ≥1.5 times baseline
  * Urine output is not included as urine could be under-captured after Foley catheter removal
Time Frame: up to approximately 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 98 | 103 | 111 | 120
Participants | 72 | 68 | 96 | 101
Statistical Analysis 1: Comparison: Lung Transplant With iNO vs Lung Transplant With iEPO; Test type: Other; p = 0.251, Chi-squared; Odds Ratio (OR) = 1.43, 95% CI 2-sided [0.78 to 2.61]
Statistical Analysis 2: Comparison: Heart Transplant & LVAD Implantation With iNO vs Heart Transplant & LVAD Implantation With iEPO; Test type: Other; p = 0.619, Chi-squared; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.58 to 2.5]

8. Secondary Outcome: Number of Participants With In-hospital Mortality
Description: Death that occurs during the hospital stay
Time Frame: up to approximately 1 year after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 98 | 103 | 111 | 120
Participants | 5 | 7 | 6 | 11

9. Secondary Outcome: Number of Participants With Post-operative Mortality Within 30 Days
Description: From the day of surgery to 30 days postoperatively.
Time Frame: up to approximately 30 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 98 | 103 | 111 | 120
Participants | 2 | 1 | 4 | 7
Statistical Analysis 1: Comparison: Lung Transplant With iNO vs Lung Transplant With iEPO; Test type: Other; p = 0.614, Fisher Exact; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.19 to 23.82]
Statistical Analysis 2: Comparison: Heart Transplant & LVAD Implantation With iNO vs Heart Transplant & LVAD Implantation With iEPO; Test type: Other; p = 0.5424, Fisher Exact; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.17 to 2.12]

10. Secondary Outcome: Number of Participants With Post-operative Mortality Within 90 Days
Description: From the day of surgery to 90 days after index surgery
Time Frame: up to approximately 90 days after index surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
Number analyzed (Participants) | 98 | 103 | 111 | 120
Participants | 4 | 4 | 5 | 12

ADVERSE EVENTS:
Time Frame: Collected from surgery to one year.
Description: Patients who were consented and randomized, but excluded or withdrawn prior to surgery and treatment are not included in this cohort description. No participant data was retained after patient exclusion or withdrawal prior to surgery and treatment. Due to the nature of the study design, comparative trial evaluating two standard of care medications, the only SAE reported is mortality at specified intervals.
Arm/Group | Lung Transplant With iNO | Lung Transplant With iEPO | Heart Transplant & LVAD Implantation With iNO | Heart Transplant & LVAD Implantation With iEPO
All-Cause Mortality (participants affected / at risk) | 9/98 | 10/103 | 10/111 | 21/120
Serious Adverse Events (participants affected / at risk) | 9/98 | 10/103 | 10/111 | 21/120
Other Adverse Events (participants affected / at risk) | 42/98 | 41/103 | 40/111 | 48/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lung Transplant With iNO (N=98) | Lung Transplant With iEPO (N=103) | Heart Transplant & LVAD Implantation With iNO (N=111) | Heart Transplant & LVAD Implantation With iEPO (N=120)
All Cause Mortality (General disorders) | 9 (9) | 10 (10) | 10 (10) | 21 (21)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lung Transplant With iNO (N=98) | Lung Transplant With iEPO (N=103) | Heart Transplant & LVAD Implantation With iNO (N=111) | Heart Transplant & LVAD Implantation With iEPO (N=120)
Venous Thromboemolic DVT (Blood and lymphatic system disorders) | 27 (27) | 21 (21) | 21 (21) | 28 (28)
Venous Thromboembolic PE (Blood and lymphatic system disorders) | 5 (5) | 10 (10) | 4 (4) | 4 (4)
Venous Thromboembolic Other (Blood and lymphatic system disorders) | 13 (13) | 10 (10) | 8 (8) | 17 (17)
Arterial Thromboembolic TIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Arterial Thromboembolic CVA/Stroke (Blood and lymphatic system disorders) | 6 (6) | 2 (2) | 7 (7) | 8 (8)
Arterial Thromboembolic Myocardial Infarction (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0)
Arterial Thromboembolic Mesenteric Ischemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Arterial Thromboembolic Other (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
LVAD Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
New Onset Atrial Fibrillation (Cardiac disorders) | 11 (11) | 18 (18) | 10 (10) | 9 (9)
Upper GI Bleed (Gastrointestinal disorders) | 2 (2) | 5 (5) | 4 (4) | 6 (6)
Lower GI Bleed (Gastrointestinal disorders) | 1 (1) | 4 (4) | 2 (2) | 6 (6)
Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/52/NCT03081052/Prot_SAP_000.pdf